CLINICAL TRIAL: NCT02424487
Title: Intracuff Pressure During One-lung Ventilation in Infants and Children
Status: Completed | Type: Observational
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chairman of department, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB14-00826
Record Dates: First submitted 2014-11-14; First posted 2015-04-23 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: One-lung Ventilation (OLV)
Keywords: Initial pressure; changes of intracuff pressure; infants and children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intracuff pressure during one-lung ventilation: Measurement of changes in intracuff pressure with one-lung ventilation during thoracic surgery.
  Interventions: Procedure: Intracuff pressure measurement in one-lung ventilation during thoracic surgery

INTERVENTIONS:
Procedure: Intracuff pressure measurement in one-lung ventilation during thoracic surgery

SUMMARY:
The purpose of this study is to evaluate the initial pressure and changes of the intracuff pressure during one-lung ventilation (OLV) in infants and children during thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients 0-18 yars old.
* Patients requiring intubation with a cuffed specialized endotracheal tube or bronchial blocker.
* Patients having thoracic surgery.
* Patients that require one-lung ventilation (OLV).

Exclusion Criteria:

* Patients that do not require to have cuffed specialized endotracheal tube or bronchial blocker.
* Patients not requiring one-lung ventilation.
* Patients not having thoracic surgery.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male and female from 0-18 years old having thoracic surgery and requiring one-lung ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-05; Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
Intracuff pressure during OLV | intraoperative
  Evaluate changes in intracuff pressure with OLV during thoracic surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Tobias, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States